CLINICAL TRIAL: NCT06322160
Title: The Role of tHyroid cAncer Specific Patient Concerns iNventory (PCI-TC) in Enhancing Shared decisiOn Making
Acronym: HANSOM
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: ENT UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 5714
Record Dates: First submitted 2024-02-06; First posted 2024-03-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No use of PCI-TC in clinical consultations: In this phase we aim to explore the views of the current decision-making process in thyroid cancer treatment. The patients will be approached for interview within 14 days after their consultations where the treatment decisions for their low risk differentiated thyroid cancer are made. There is no time restriction to approach clinicians for interview.
  Interventions: Other: Interview
- User experience of PCI-TC in thyroid cancer outpatient clinic setting: First, the clinicians will be trained on how to use the PCI-TC in their outpatient clinics. A new group of patients will then be identified and recruited for the phase two study. Patients from this new group will be given the PCI-TC in a quiet area just off the waiting area prior to the consultation. They will be asked to tick items on the PCI-TC list which they wish to discuss. The clinicians will conduct the consultation using the ticked PCI-TC as a guide and discuss with patients regarding the treatment plan for their thyroid cancer. The patients will be approached for interview within 14 days after their consultations. The clinicians will be approached for interview after all recruited patients in phase two study have had their consultation regarding their cancer treatment.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Interview with individual participant will take place via online videoconferencing MS Teams

SUMMARY:
Multiple clinical equipoises exist for the management of thyroid cancers. Shared decision-making (SDM) process where patients are supported to consider options, to achieve informed preferences with their clinicians have been recommended to improve patients' satisfaction and their overall quality of life. However, SDM can be difficult to achieve in our standard clinical encounters due to clinician's lack of confidence and time limitation to elicit patient's concerns and preferences. PCI as a decision-making support tool has shown to enhances clinician's awareness of patient's needs and allows for a more effective communication while the consultation time is unaffected. The successful development, testing and implementation of a PCI-TC could improve patient satisfaction, clinical efficiency and ensure that unmet need is appropriately addressed. This study will support the development of PCI-TC to better understand the wide-ranging needs of our patients and to improve the SDM process in the thyroid cancer management pathway.

DETAILED DESCRIPTION:
Differentiated thyroid carcinoma (DTC) is currently one of the most rapidly increasing tumours. And it is predicted to continue to rise over the next 10 years (1). Surgery to remove the entire thyroid gland remains the gold standard treatment for low-risk DTC with (tumour size between 1cm to 4cm). The extent of thyroid resection for low-risk disease however is controversial. Until recently, the standard of care has been a 'one size fits all' approach of total-thyroidectomy (TT) for >1cm DTC. This treatment has afforded excellent overall survival rate (98-99% at 10-year) and a low recurrence rate (2-8% at 7-year) (2). However, based on recent studies, national guidelines (American Thyroid Association 2015 and British Thyroid Association 2014) now propose hemithyroidectomy (HT) as potentially adequate treatment in low-risk DTC (3,4). This is because TT does not appear to offer an overall survival advantage over HT, and subject patients to life-long hormone replacement therapy and perhaps an increased risk of postoperative complications. However, the recent change in guidance is only based on retrospective and observational single-centre studies which are subject to various types of bias (5). A clear "surgical equipoise" therefor exists for managing low-risk thyroid cancer patients. When faced with this equipoise, where clinicians are not sure and data are still equivocal, it is even more difficult for patients to understand the issues and make a treatment choice that is best for their individual needs and priorities. Due to the excellent prognosis, there is an ever-increasing pool of cancer-survivors in whom long-term quality-of-life (QoL) is more important than cure rates. Many thyroid cancer patients have severe anxiety and long-term problems resulting in low QoL. Unfortunately, a recent National Patient Survey showed that existing clinical equipoise (and resulting practice variation) has resulted in high levels of confusion, dissatisfaction, and anxiety in patients with regards to treatment decision (6). Enabling better patient decision-making to choose the best treatment choice should lead to an improved patient experience, higher satisfaction, better QoL and reduced health burden on the NHS (7).

Patient concerns inventory (PCI) is a condition-specific prompt list which allows patient to formulate an individualised record of their concerns, needs and priorities that can be used as a structure to help guide out-patient consultations (8). Patients identify, in advance of consultations, salient issues from a specifically designed questionnaire prompt list (PCI). This allows clinicians to focus dialogue quickly on patients' main concerns and to address issues that patients might be otherwise have been reluctant to discuss. The original PCI was developed by Professor Simon Rogers, consultant oral and maxillofacial surgeon of Aintree University Hospital, Liverpool, in 2009 to provide a patient focused approach to managing head and neck cancer (8). Since then, PCIs have also been successfully developed in other disciplines such as breast cancer (9), burns (10), rheumatology (11), stroke care and diabetes.

Recently we have developed a thyroid-specific patient concerns inventory (PCI-TC) [see Appendix for Thyroid Concerns Inventory] from literature review on the unmet needs of thyroid cancer patients followed by two phases and six rounds of modified Delphi process within a thyroid cancer multi-disciplinary team (MDT). We hope the use of PCI-TC at diagnosis will help tease out patient's top concerns and expectations regarding their treatment and care going forward, thus enhancing shared decision making (SDM), so that they are better informed and have confidence in their treatment preferences/choices within the current equipoise.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Both genders
* Patients who are diagnosed of low-risk well-differentiated thyroid carcinoma (papillary thyroid carcinoma or follicular carcinoma) with size of 1-4cm. This is either:

  1. Diagnosed pre-operatively by fine-needle aspiration cytology (FNAC) with Thy5 grade [see appendix for the Thy classification] or
  2. Confirmed following diagnostic hemithyroidectomy
* Able to communicate in spoken and written English

Inclusion criteria for clinician participants

* Consultant head and neck and thyroid surgeons who directly involve in the diagnosis and/or management of low-risk well-differentiated thyroid cancer (papillary thyroid carcinoma or follicular carcinoma) with size of 1-4cm for at least ten patients per year.
* Both genders
* Able to communicate in spoken and written English

Exclusion Criteria:

* Patients who are diagnosed with tumour with adverse features this includes:

  * Tumour with poor differentiated cytology or variants with bad prognosis (tall cell, columnar cell, Hurthle cell, solid variant)
  * Tumour, which is multifocal, bilateral, with extrathyroidal extension, with perineural or lymphovascular invasion.
  * Tumour with clinically or radiologically involved nodes or distant metastases
  * Tumour which is of a familial disease
* Patient who is either Pregnant or breast-feeding
* Patient with hyper- or hypothyroidism who is a candidate for surgery
* Patient who is concurrently diagnosed with any medullary, anaplastic, lymphoma, or parathyroid disease
* Patients who had previous thyroidectomy for reasons other than diagnostic hemithyroidectomy for their recent cancer diagnosis.
* Patients who are cognitively impaired or have a mental health condition and are therefore unable to give consent
* Patient who is not able to read write and speak English.

Exclusion criteria for clinician participants

• Consultant surgeons who diagnose and/or manage low-risk well-differentiated thyroid cancer for less than ten patients per year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We also aim to include 4 consultants head and neck and thyroid surgeons in the study centres.
  Patients who have been diagnosed with low risk differentiated thyroid carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
To explore patients' and clinicians' view and experience of the current decision-making process for low risk differentiated thyroid cancer | through study completion, an average of 1 year
  • To explore clinicians' and patients' user experience of thyroid cancer specific patient concerns inventory (PCI-TC) in thyroid cancer outpatient clinics through the interviews conducted. Qualitative study rather than assessment.
• To explore clinicians' and patients' user experience of thyroid cancer specific patient concerns inventory (PCI-TC) in thyroid cancer outpatient clinics. | End of study
  • To explore clinicians' and patients' user experience of thyroid cancer specific patient concerns inventory (PCI-TC) in thyroid cancer outpatient clinics.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Guys & St Thomas, London
  - UCLH, London

IPD SHARING:
Plan to Share IPD: No